Study Title: P50 Pragmatic Implementation Science Approaches to Assess and Enhance Value

of Cancer Prevention and Control in Rural Primary Care

Principal Investigator: Russell Glasgow

COMIRB No: 19-1706 Version Date: 04/22/21

You are being asked to be in this research study because you are between 55-80 years of age and a current smoker or quit smoking in the last 15 years.

If you join the study, you will be asked to complete 2 surveys. In addition, the study team will record the following information from your healthcare provider's records: your age, smoking status, smoking history, insurance status, current lung cancer symptoms (if any), current related illnesses (if any), and current smoking cessation medications (if any). All the collected information will be de-identified, which means it will be labeled only with a study subject number and not associated with your name or any identifiable information. You will be reimbursed with a \$100 gift card for your time.

This study is designed to find out if targeted education of primary care teams and informational tools can help better follow the recommendations of the US Preventive Services Task Force.

Participation in this study is completely voluntary. You do not have to be in this study if you do not want to be. If there is a question on the survey you do not want to answer, you can simply skip it. There may be risks of which the researchers may not have thought.

We will share only de-identified data in a form of summaries where no individual record can be tracked.

This research is being paid for by a grant from the National Cancer Institute.

If you have questions, you can email or call Bryan Ford at bryan.ford@cuanschutz.edu or 303.724.3422. You can call and ask questions at any time.

You may have questions about your rights as someone in this study. If you have questions, you can call the COMIRB (the responsible Institutional Review Board). Their number is (303) 724-1055.